CLINICAL TRIAL: NCT00268073
Title: Comparison of the Incidence of Neo-Aortic Insufficiency After Classic Norwood I and Norwood I-Sano Procedures
Brief Title: Incidence of Neo-Aortic Insufficiency
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-067
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: Pediatric; cardiac; neo-aortic insufficience; Norwood standard Stage I procedure; Norwood Sano procedure
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The records of all the patients that underwent the Norwood-Sano operation at Children's Healthcare of Atlanta, Emory University between January 1, 2002 and December 31, 2004 will be investigated. These patients will be compared with an equal number of consecutive cases treated by classic Norwood stage I operation in order to determine the incidence of neo-aortic valve insufficiency and the clinical outcome of these patients.

DETAILED DESCRIPTION:
Neoaortic valve insufficiency after Norwood type palliation of single ventricle patients has not been well studied. Patients with mild insufficiency tolerate it well; moderate to severe insufficiency however is poorly tolerated and can result in the death of the patient or at least require re-operation. Re-operation for neo-aortic insufficiency in this small size child is a difficult operation and the operative options are very limited. The introduction of the Sano modification of the Norwood procedure introduced a new set of variables due to the presence of a ventricular incision and possible distortion of the neo-aortic valve. It is therefore critical to determine the incidence of neo-aortic insufficiency and compare it to the standard Norwood operation, as well as to determine the clinical consequences of the presence of this phenomenon immediately postoperatively as well as long-term, up to completion of the stage II of the Norwood procedure (Glenn stage).

ELIGIBILITY:
Inclusion Criteria:

* patients undergone Norwood-Sano at Children's Healthcare of Atlanta between 9.2.2002 and 12.31.2004
* equal number of consecutive patients undergone Norwood classic stage I at Children's Healthcare of Atlanta between 9.2.2002 and 12.31.2004

Exclusion Criteria:

* those who do not meet the inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2002-01

CONTACTS AND LOCATIONS:
Overall Officials: Kirk R Kanter, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States